CLINICAL TRIAL: NCT06266195
Title: Spectroscopic Profiling of Extracellular Vesicles By Resonant Gold Nanostructures in the Infrared
Acronym: PROVEIR_1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5452
Record Dates: First submitted 2023-07-21; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-04

CONDITIONS: Vesicle
Keywords: MICROVESCICLES; CIRRHOSIS; HCC; NANOSTRUCTURES.
MeSH Terms: conditions — Blister; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GRUPPO CIRROSI: 32 soggetti uomini o donne, >18 anni con diagnosi di cirrosi epatica di differente eziologiA
  Interventions: Diagnostic Test: sierological test
- GRUPPO HCC: 32 pazienti uomini o donne, con diagnosi di neoplasia primitiva del fegato
  Interventions: Diagnostic Test: sierological test

INTERVENTIONS:
Diagnostic Test: sierological test — sierological test: circulant vescicles

SUMMARY:
Extracellular vesicles, due to their ease of extraction and ability to represent the cells from which they originate, have high potential in the field of personalized medicine, especially in the identification of new early bio-markers of cancer, including hepatocellular carcinoma. Nevertheless, the development of high-throughput diagnostic methods in this area is still in its infancy, and the design of new integrated technological solutions is of great interest and topicality. The main hypothesis of this study is that the development of a novel technology integrating resonant gold nanostructures in the mid-infrared can significantly contribute to the development of new approaches for the diagnosis of hepatocellular carcinoma.

ELIGIBILITY:
Inclusion

* 18 years old with a diagnosis of liver cirrhosis of different etiology
* 18 years old with a diagnosis of hepatocellular carcinoma

Exclusion

* Have not signed the informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of this study is divided into two groups: a) control group, 32 cirrhotic patients and b) oncology group, 32 patients diagnosed with hepatocellular carcinoma
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
primary endpoint | 12 months
  To evaluate the change in extracellular vesicle concentration between the control group and oncology group. The concentration of vesicles per ml of blood will be measured by frequency shift of the plasmonic resonance peak of gold nanostructures following immuno-capture of vesicles.

CONTACTS AND LOCATIONS:
Overall Officials: FABRIZIO PIZZOLANTE, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- FPGemelliIRCCS, Rome, Lazio, Italy